CLINICAL TRIAL: NCT05128877
Title: The Effectiveness of Relaxation Training on Primary Dysmenoreh and Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emir İbrahim IŞIK, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PrimDys01
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Menstrual Discomfort; Relaxation Abnormality; Dysmenorrhea Primary
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental study.
Who Masked: Participant
Masking Description: The women included in the study will be divided into 2 groups as experimental and control groups by applying randomization using the random drawing method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention was made in the control group.
- intervention group (Experimental): Progressive relaxation techniques were applied to the intervention group.
  Interventions: Other: relaxation techniques

INTERVENTIONS:
Other: relaxation techniques — Mitchell's physiological relaxation technique is based on reciprocal inhibition and involves diaphragmatic breathing and a series of ordered isotonic contractions.
  Arms: intervention group

SUMMARY:
The aim of this study is to evaluate the effectiveness of Laura Mitchell's relaxation training on primary dysmenorrhea and menstrual symptoms. The study will be carried out on women who have been diagnosed with primary dysmenorrhea, have a regular menstrual cycle (28±7 days), have menstrual pain higher than 4 cm according to the visual analog scale (VAS), and wish to voluntarily participate in the study. The questionnaire created by the researchers will be administered online. The women included in the study will be divided into 2 groups as experimental and control groups by applying randomization using the random drawing method. Laura Mitchell's physiological relaxation training will be applied to the experimental group for 30 minutes on menstrual days during a total of 3 menstrual cycles, accompanied by an online live lesson. The control group will continue their daily routine.

DETAILED DESCRIPTION:
Dysmenorrhea is a common gynecological complaint in women of reproductive age, characterized by lower abdominal pain that occurs a few hours before or with the onset of menstruation and persists for 1-2 days. It is more common in adolescent and young women. It is divided into primary and secondary dysmenorrhea. The prevalence of primary dysmenorrhea varies between 17-95%. Primary dysmenorrhea, unlike secondary dysmenorrhea, is due to contraction of the myometrium without pelvic pathology. Pain occurs with every menstrual cycle. Generally, cramp-like pain in the suprapubic region may be accompanied by nausea, vomiting, headache, dizziness, sweating, diarrhea, insomnia and syncope . While primary dysmenorrhea is more common in nulliparous, both its severity and incidence decrease with increasing age and parity. Primary dysmenorrhea is pelvic pain that is caused by the natural production of prostaglandins and is not associated with pelvic pathology, and is among the common causes of admission to emergency services. In the pathogenesis of primary dysmenorrhea, it is thought to be associated with prostaglandin production, which increases with vasoconstriction of the uterine blood vessels, leading to uterine contractility and ischemia. Primary dysmenorrhea does not threaten the life of women, but it can affect the quality of life negatively and prevent work and school continuity. There are various relaxation techniques in the literature to reduce the pain and improve the quality of life of women with primary dysmenorrhea. Relaxation techniques are effective and easy-to-apply self-management therapy in reducing the effects of pain, stress, depression, anxiety and mood changes on the individual and in controlling the body. Laura Mitchell's Simple Physiological Relaxation Training is a standard method with the advantages of requiring less concentration, being learned in a short time and showing a rapid effect, and is widely used especially in the field of obstetrics and gynecology. It is known that this technique, which includes diaphragmatic breathing, improves immune system functions and quality of life, and also reduces depression. The aim of this study is to evaluate the effectiveness of Laura Mitchell's relaxation training on primary dysmenorrhea and menstrual symptoms.

METHOD The study will be carried out on women who have been diagnosed with primary dysmenorrhea, have a regular menstrual cycle (28±7 days), have menstrual pain higher than 4 cm according to the visual analog scale (VAS), and wish to voluntarily participate in the study. The questionnaire created by the researchers will be administered online. Before starting the study, the consent of the participants will be obtained via online link. The women included in the study will be divided into 2 groups as experimental and control groups by applying randomization using the random drawing method. Data collection Evaluations were evaluated according to the physical (age, height, body weight, body mass index) and demographic data of the individuals (age at menarche, mean cycle duration, duration of menstruation, pain status, duration of pain, number of pads used on the busiest day, presence of menstrual symptoms experienced during menstruation period). intensity) will be recorded. Individuals will be examined for 5 menstrual cycle follow-ups, 4 of which are consecutive. Pain intensity of individuals will be evaluated with Visual Analog Scale (VAS) and menstrual symptoms will be evaluated with Menstrual Symptom Scale (MSS). To the individuals participating in our study; The 1st day of the 1st menstruation is the 1st evaluation, and the data will be collected with VAS and MSS for both groups, and relaxation training will begin for the experimental group. The 1st day of the 2nd menstruation is the 2nd evaluation, and the data will be collected with VAS and MSS for both groups, and relaxation training will be continued for the experimental group. The 1st day of the 3rd menstruation will be the 3rd evaluation. Data will be collected with VAS and MSS for both groups, and relaxation training will be continued for the experimental group. The 1st day of the 4th menstruation will be the 4th evaluation, and the data will be collected with VAS and MSS for both groups, and the relaxation training will be terminated for the experimental group. They will be free to continue exercising until the seventh menstruation. 1st day of 7th menstruation

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary dysmenorrhea, have a regular menstrual cycle (28±7 days), menstrual pain greater than 4 cm on the visual analog scale (VAS) women willing to participate in the study voluntarily

Exclusion Criteria:

* Gastrointestinal, urogynecological, autoimmune, psychiatric diseases, other chronic pain syndromes, childbirth, positive pregnancy test, breastfeeding, intrauterine device users, pelvic surgery users, using chronic medication, including oral contraceptives or antidepressants for at least 6 months before the study, irregular menstrual cycle women (with a cycle duration of less than 21 days or longer than 35 days) and women with a pathological history or ultrasonographic imaging showing secondary dysmenorrhea

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 months
  for pain

SECONDARY OUTCOMES:
menstrual symptom questionnaire | 6 months
  for menstrual symptom discomforts

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided